CLINICAL TRIAL: NCT01233700
Title: Brief Nursing Intervention to Prevent Poor Psychosocial Outcomes in Living Donors
Brief Title: Brief Intervention to Prevent Poor Psychosocial Outcomes in Living Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mary Amanda Dew, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21NR011149 (NIH); R21NR011149 (NIH)
Record Dates: First submitted 2010-10-26; First posted 2010-11-03 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Living Donation
Keywords: living donation; organ donation; psychological adaptation; mental health; physical well-being; interpersonal relations; quality of life; psychosocial factors
MeSH Terms: conditions — Psychological Well-Being | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motivational Interviewing (Experimental): Subjects will receive two, individual telephone sessions with an interventionist, each lasting approximately 30-45 minutes. The sessions will focus on assisting subjects to delineate their reasons for or against proceeding with living organ donation and assisting subjects to resolve any lingering concerns about their decisions regarding donation.
  Interventions: Behavioral: Motivational Interviewing
- Enhanced Standard Care (Active Comparator): Subjects will receive two individual telephone sessions with an interventionist, each lasting approximately 30-45 minutes. The sessions will focus on providing educational information to subjects regarding healthy lifestyle issues (healthy eating, diet, exercise, quitting smoking).
  Interventions: Behavioral: Healthy Lifestyles Education
- Standard Care (No Intervention): Subjects will receive the standard care and education provided by the Living Donor Program at their medical center.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Standard motivational interviewing techniques will be applied to assist subjects to consider and work to resolve any remaining concerns, doubts, or ambivalence about their decision about donating an organ to someone else.
  Arms: Motivational Interviewing
Behavioral: Healthy Lifestyles Education — Educational information will be presented to subjects in didactic form on lifestyles issues of relevance to living donors.
  Arms: Enhanced Standard Care

SUMMARY:
The purpose of this study is to evaluate the potential effectiveness of a psychosocial intervention based on the principles of motivational interviewing. The novel intervention will assist living donor candidates to think through any remaining concerns or questions that they may have about living donation. If the intervention is effective, it may help to prevent post-donation problems related to psychological and health outcomes.

DETAILED DESCRIPTION:
The protection of living donors' well-being and the prevention of any negative consequences of donation are among the foremost priorities in transplantation. Some donors experience poor psychosocial outcomes after donation, including psychological distress, poor perceived physical well-being, and strained family relationships. No preventive interventions have been mounted or tested for their ability to avert poor psychosocial outcomes in living donors. The present study will provide an initial test of a new intervention for this purpose. The new intervention utilizes motivational interviewing (MI) to address remaining concerns that individuals may have about proceeding with living donation. Study participants will be randomly assigned to either (a) participate in the MI intervention (during which they will be asked to answer a series of questions to help them better delineate their reasons for and against proceeding with living organ donation), (b) participate in a comparison intervention designed to inform them about healthy lifestyle habits, or (c) not receive any intervention. We plan to recruit a maximum of 150 adults who are considering whether to serve as living kidney or liver donors. We hypothesize that participants receiving the MI intervention will have superior outcomes (less psychological distress, fewer physical health complaints, better interpersonal relationships within their family, better overall quality of life)after donation.

ELIGIBILITY:
Inclusion Criteria:

* Score of 1 or greater on the Simmons Ambivalence Scale;
* Must be able to speak English;
* Have been evaluated as a potential living kidney or liver donor candidate;
* Aged 18 or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
psychological distress | 6 weeks post-donation
  PRIME-MD depression and anxiety modules, Brief Symptom Inventory (BSI) anxiety items, Simmons Feelings About Donation items; Simmons Psychosocial Concerns About Donation items
somatic/physical health perceptions | 6 weeks post-donation
  Concerns About Donation Effects items, Simmons Post-donation Medical Concerns, Brief Pain Inventory short form, FACIT-fatigue scale, Post-surgery Body Image Questionnaire, Post-donation Symptom Checklist, Simmons Concerns About Future Health items, Simmons Perceived Stressfulness of Donation items
interpersonal relationship quality and distress | 6 weeks post-donation
  Simmons Family Relationship items, Short Dyadic Adjustment Scale, Family ICPS conflict and intimacy subscales
quality of life | 6 weeks post-donation
  RAND-12
psychological distress | 3 months post-donation
  PRIME-MD depression and anxiety modules, BSI anxiety items, Simmons Feelings About Donation items; Simmons Psychosocial Concerns About Donation items
somatic/physical health perceptions | 3 months post-donation
  Concerns About Donation Effects items, Simmons Post-donation Medical Concerns, Brief Pain Inventory short form, FACIT-fatigue scale, Post-surgery Body Image Questionnaire, Post-donation Symptom Checklist, Simmons Concerns About Future Health items, Simmons Perceived Stressfulness of Donation items
interpersonal relationship quality and distress | 3 months post-donation
  Simmons Family Relationship items, Short Dyadic Adjustment Scale, Family ICPS conflict and intimacy subscales
quality of life | 3 months post-donation
  RAND-12

SECONDARY OUTCOMES:
Satisfaction with intervention | pre-donation (on average, 1 week post-intervention but before donation has occurred)
  adapted Client Satisfaction Scale
Quality of decision to donate | pre-donation (on average, 1 week post-intervention but before donation has occurred)
  Simmons Ambivalence Scale items; Decision Conflict Scale, Decision Satisfaction Scale items

CONTACTS AND LOCATIONS:
Overall Officials: Mary Amanda Dew, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Dew MA, DiMartini AF, DeVito Dabbs AJ, Zuckoff A, Tan HP, McNulty ML, Switzer GE, Fox KR, Greenhouse JB, Humar A. Preventive intervention for living donor psychosocial outcomes: feasibility and efficacy in a randomized controlled trial. Am J Transplant. 2013 Oct;13(10):2672-84. doi: 10.1111/ajt.12393. Epub 2013 Aug 7. PMID 23924065